CLINICAL TRIAL: NCT00749645
Title: Clinical Phase II Pilot Study of the Efficacy of FANG(30) to Treat Active Rheumatoid Arthritis in Adult Patients
Brief Title: Efficacy Study of FANG(30) for Active Rheumatoid Arthritis in Adult Patients
Acronym: FANG30-RA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Juan C. Bertoglio, MD (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Sponsor-Investigator, Juan C. Bertoglio, MD, Principal Investigator, Universidad Austral de Chile
Organization: Universidad Austral de Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCT06-AG-02; DO4I1240FONDEF (Other: CHILE Scientific Technological Development Fund)
Record Dates: First submitted 2008-09-07; First posted 2008-09-09 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2014-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid, Andrographolides treatment, Efficacy.
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - FANG(30) (Active Comparator): 1 - Active comparator, consisted of 30 adult patients with active Rheumatoid Arthritis, randomly assigned, taking the active product, in addition to base medication (Mtx + Pdn)
  Interventions: Drug: FANG(30)
- 2 - Placebo (Placebo Comparator): 2 - Placebo comparator, consisted of 30 adult patients with active Rheumatoid Arthritis, randomly assigned, taking the placebo formulation, in addition to base medication (Mtx + Pdn)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FANG(30) — Andrographolide formula Oral tablets, 30mg, three times per day, during a total of 105 continuous days.
  Other Names: FANG 30mg tablets, FARMINDUSTRIA, Lots FANG06 & 01-ANDRO-07
  Arms: 1 - FANG(30)
Drug: Placebo — Placebo 30mg tabs, 3/day, 105 days continuously.
  Other Names: FARMINDUSTRIA Specific Placebo tabs/Lot FANG06 & 01-ANDRO-07
  Arms: 2 - Placebo

SUMMARY:
This is a Clinical Pilot Phase II interventional, double blind, randomized and placebo controlled study to document the efficacy, tolerability and safety of FANG(30) in 60 adult patients affected with active Rheumatoid Arthritis. Also, to evaluate the effect of an andrographolide natural formula, identified as FANG(30) or "the study product", on the immunological functions that influence chronic inflammatory process in these patients, who could benefit with this treatment.

DETAILED DESCRIPTION:
Introduction: Rheumatoid Arthritis (RA) is a common rheumatic disease characterized by pain, inflammation and reduction in joint function. Hands and feet are the most commonly affected joints and pain is the cause that brings patients with RA to search for medical assistance. Factors causing pain and the risk of physical incapacity are still poorly understood. Joint pain in RA is, generally, a profound pain, focalized in the involved joint. Typically, pain increases when joint moves and decreases when joint is at rest. But, in the advanced form of the disease, pain can be persistent and some patients can feel night pain, or rigidity and pain after a period of inactivity, that last more than 1 hour and decreases when some activity is taken up again, i.e. rigidity and early morning pain. Clinically, these patients present with symptoms such as localized sensibility on the joints, and slight edema of the tissue, bone crepitating and heat on the outer joint. Muscular atrophy with or without muscular spasm can be seen. In the advanced form of the disease, there is deformity and complete loss of joint movement. Analgesic drugs, specially the non steroidal anti-inflammatory drugs NSAIDs play an essential role in the management of RA. These drugs are not only effective in the rapid and sustained relief of pain, but at the same time they can have an acceptable profile of safety and tolerability in medium and long term treatment. However, there are cases of gastric intolerance and /or renal or hepatic dysfunction. The anti-inflammatory effect of non steroidal anti-inflammatory drugs NSAIDs, is mainly due to the inhibition of the cyclooxygenase enzyme (COX), that is needed for the synthesis of prostaglandins and thromboxanes.

Description of FANG used in this clinical trial: FANG(30) is a product manufactured by FARMINDUSTRIA S.A., Pharmaceutical Laboratories, Santiago, Chile, in the form of a common medicine, according to Good Manufacturing Practices (GMP) Guidelines & Requirements of the Institute of Public Health of Chile (ISP), from a standardized and patented extract of A. paniculata, Nees (Acanthaceae), a medicinal plant native to India and China. Its chemical composition and principal active compounds are bitter diterpenic lactones, specially andrographolide, deoxy-andrographolide and neoandrographolide, in tablets weighting 100 mg with a 30 % of the active principle. This plant is vastly distributed in the countries of Southeast Asia and has been used as an official medicinal plant in China and India for thousands of years. It still continues as a popular medicine for the treatment of different diseases. Recently it has been demonstrated to possess anti tumoral5, anti-inflammatory6 and antiviral7 effects. Andrographolide is particularly efficient in regulating the immune response 5, 7. The molecular and cellular mechanisms responsible for the immunomodulating and anti-inflammatory properties of andrographolide, remain still unknown, however, recent in vitro and in vivo studies, indicate that andrographolide inhibits NFkappaB8. Specifically, andrographolide in concentrations of 10 µM interferes with the DNA binding of NF-κB reducing the expression of COX-2 in neutrophils induced with fMLP and PAF. Moreover, andrographolide reduces the production of IFNγ and IL-2 in T cells stimulated with CON-A, without affecting the cellular viability or inducing apoptosis. Also the apoptosis induced by corticosteroids in thymocytes was reduced. Andrographolide and 14-deoxyandrographolide are able to inhibit the ERK1/2 phosphorylation in T cells and neutrophils, respectively 9, 10. In inflammatory processes, FANG has shown potent anti-inflammatory effects, reducing the production of cytokines, derived from phospholipids, nitric oxide and reactive oxygen species that are the "fuel" for chronic inflammation, explaining its capacity to reduce and control inflammation, inflammatory pain and facilitate the induction of cellular repair. Clinical Evidence of some effects of A. paniculata: During the last decades, A. paniculata has become popular in Scandinavia for the treatment of common cold. Accumulated evidence indicates that it can reduce the severity of this disease. Various clinical studies indicate that A. paniculata is effective for the treatment of viral infections of the upper respiratory tract. A meta-analysis in 2004 on 7 double blind controlled clinical trials that met the criteria and scientific quality accepted for this meta design, including 896 participants, which evaluated the efficacy of A. paniculata for the treatment of acute respiratory infections11, indicates in the combined results, that A. paniculata was more effective than the placebo in reducing the symptoms of common cold. A. paniculata has also been compared to acetaminophen. In a double blind randomized study with 152 patients with fever and pharyngeal congestion 12 high doses of A. paniculata (6 g) reduced fever and sore throat in a similar manner to acetaminophen, without significant secondary effects. In a double blind randomized trial, against a placebo, with 107 patients, A. paniculata increased resistance to common cold 13, reducing the incidence of colds by a factor of 2.1 times compared to the control group after a 3 months treatment during winter season. Safety Parameters - Toxicity and Tolerability of FANG: Acute and sub-chronic toxicity in rodents and pigs using an extract of A. paniculata the component of FANG, performed at the Institute of Pharmacology and Toxicology, Universidad Austral de Chile according to Good Laboratory Practice (GLP) and Food Administration Agency (FDA), showed the absence of adverse effects with doses >20g/kg after 90 days of treatment. Not genetic, or reproductive, immunological, neurological, hematological, metabolic, histopathological toxicity were detected either. Also, in a Phase I clinical trial, where the participants were monitored for liver, renal and hematological parameters, no clinical or laboratory secondary effects were described 11, 13, 15. Bio safety studies in small children, nursing mothers, patients with renal or hepatic damage have not been performed yet. On the other hand, since A. paniculata can stimulate the contractibility of gall bladder. Therefore, it should not be used without medical supervision or in patients with gall bladder pathology.

Objective of Study: To assess and measure the anti inflammatory efficacy of this test natural product and contribute learning about some of the basic biological mechanisms by which produces its effects, on adult patients with active Rheumatoid Arthritis. Methodology: For this purpose, there will be 2 groups of patients who will respectively receive at random, an either inert substance known as placebo, and the other group that will receive the test product in the form of coated tablets, three times every day, during the period of study that will last 14 weeks.

Place of Study: National study in Chile with 2 centers, one in the city of Valdivia and one in the city of Osorno with a number of 30 patients per centre and enrolled by their respective rheumatologists. Population of Study: 60 adult individuals of both sexes diagnosed with Active Rheumatoid Arthritis and undergoing standard treatment will be included. Individuals with chronic or acute disease, smokers, alcoholics, diabetics, heart diseases, lung diseases, neoplastic diseases, and individuals taken any other medicine will be excluded. Product of Study: The experimental FANG (30) and the placebo tablets were manufactured and stored as specified, and will be delivered and administered as proposed in this protocol. Procedure: A total of approximately 30 individuals will be assigned to the placebo group, and 30 to the FANG(30) group. During 14 weeks, each of them will daily take 3 tablets of the respective randomly assigned product. All volunteers will allow obtaining a monthly blood sample by simple venipuncture from the superior arm at day 0, 30, 60, 90 and 120 days of treatment.

Discomfort and derived risks of the study: Since the participants, will need to take tablets of the product 3 times a day and submitted to the extraction of 4 blood samples during the study period, these facts can represent in some cases, a physical and emotional discomfort, depending of the customs and individual predisposition for this type of common medical procedures. Adverse Effects: Andrographis paniculata extract is not toxic and the manufactured product FANG(30) is prepared under GMP with pharmaceutical quality as requested for this study. The product is well tolerated and no complications are reported in the vast available information. However, as any natural and / or pharmaceutical product, in isolated cases, there can be slight risks such as rushes, allergies to the active principles of the plant, which anyhow, are reversible with the suspension of the intake of the product. Moreover, if in one of the patients, an alteration is detected that could be dangerous or inconvenient for his or her health condition; physicians will offer this patient to withdraw from the study. In case of a severe alteration, the rheumatologist will withdraw the patient from the study for safety reasons.

Principal expected results: At the end of the study period, participants receiving the active product FANG (30) (Andrographis extract tablets), should show an improvement in their symptoms. Moreover, participants that received placebo should not show any sign of change in their symptoms. Any situation of health detected during the course of the study, related to the analyzed parameters, or any other aspects of clinical significance, even not necessarily included in this study, will be duly recorded and informed accordingly. If end results demonstrate that FANG(30) in a particular case has proven to be beneficial, all participating patients (even those having received a placebo) will be offered by their rheumatologists a free treatment with this same medicine in a regular modality, for the next 18 months.

Volunteering: Volunteers must be absolutely free to apply and participate, in order to be included in this study, as for no reason whatsoever nobody can oblige a person to participate under any condition or threat. Moreover, volunteers can abandon and not continue participating in this study at any moment and without necessity of given explanations. This event will not affect the relationships with treating physicians, neither with the personnel of the hospital, or have any relation or influence with volunteer's future health care requirements. Volunteers can, and must consult all doubts about the study in which they have been invited to participate, before accepting and also during development of the study. Insurance for the Study: Considering the previous experience with the drug, of being of free sale in other countries; being approved by the Institute of Public Health in Chile, authorized to be sold as a nutraceutical in the USA, no hiring of specific insurance for special risks of this study has been considered. Moreover, this study has no special funds for the payment of compensations for damages resulting from adverse effects to the test medicine. Nevertheless, in case some event of this nature would happen, volunteers will be assisted with all the procedures and therapies they require, and continue to be monitored by a study physician for their care. In case of additional interventions needed, but not derived directly from adverse effects of this study and not covered by regular health insurance systems, these events will be also covered by the insurance policy of this study. This insurance policy will be maintained current for up to 4 months after the completion of the study. Responsible rheumatologists to inform volunteers on the study, to clarify doubts or answering questions are Dr. Verónica I. Aguirre at Hospital de Valdivia and Dr. Sonia M. Arriagada at Hospital de Osorno.

ELIGIBILITY:
Inclusion Criteria:

* Patients, between 18 and 70 years of age.
* Clinical diagnosis of RA, based on typical history and clinical presentation of the patient according to the diagnostic criteria of the American College of Rheumatology (ACR), 1987.
* Active AR characterized by pain and increase in joint volume, in at least 1 joint, associated to VHS > 20 mm/h and/or PCR > 0,6 ng/ml.
* Ambulatory patient requiring treatment with anti-inflammatory drugs, whom is neither receiving non-steroidal anti-inflammatory drugs (NSAIDs) nor any other drugs, except Paracetamol, for at least 4 weeks previous to the beginning of the study.
* Also, patients with RA treated with Prednisone and/or Chloroquine and Methotrexate in stable doses for at least 6 weeks, with active arthritis, and willing to participate in the study.
* Willing to come to regular controls.
* Written consent signed by the patient, according to the criteria and text approved by the local Scientific Ethical Committee.

Exclusion Criteria:

* Pregnant women, breast feeding, childbirth, potentially fertile and / or not following adequate contraceptive methods.
* Non degenerative joint diseases or other joint diseases that could interfere with the evaluation of RA (i.e. Gout, Pseudogout, Chondrocalcinosis, Psoriatic Arthritis, Infectious Arthritis, Reactive Arthritis or Spondylitic Arthritis).
* Severe disabling arthritis leaving the patient eligible for surgical intervention, or incapacitated and prostrated patients.
* Treatment with intra-joint injection with corticosteroids one month before treatment.
* Ongoing treatment with anticoagulants, hydantoins or lithium.
* Presence or history of digestive hemorrhage, peptic ulcer in the 6 previous months or hemorrhagic ulcer any time during the past, gall bladder stones or dysfunction.
* Hypersensitivity and / or intolerant to NSAIDs, including patients with bronchospam history induced by Aspirin.
* Evidence of renal, hepatic and severe hematopoietic diseases, and heart failure revealed by laboratory tests or other tests.
* History of using any other test drug, one month before to the beginning of this trial.
* Patients with tranquilizers, hypnotic or excess of alcohol, which can interfere with the perception of pain.
* Necessity of any other therapy for arthrosis, except Paracetamol used as a rescue drug during the period of study. Also exercise and/or physiotherapy, if ongoing, can continue without modification.
* Not willing to come for regular follow ups during the period of duration of the study.
* Non cooperative attitude.
* Any condition that in the opinion of the physician, does not justify the inclusion of the patient in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-10; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Primary: Day1, end of week2, then every 4 weeks for 105 days, the following will be measured: 1.Inflamed and painful joints count. 2. Intensity of pain by patient on Visual Analogue Scale(VAS). 3. Overall improvement by HAQ and SF 36 (enclosed). | Monthly

SECONDARY OUTCOMES:
Secondary:Day1, end of week2, then every 4 weeks for 3 mo, it will be measured: Morning stiffness duration. | Monthly
Symptoms relief by patient and researcher. | Monthly
Paracetamol used as rescue medicine for pain. | Monthly
Tolerability by patient and researcher. | Monthly

CONTACTS AND LOCATIONS:
Overall Officials: Juan L. Hancke, DVM, PhD, Study Chair — Universidad Austral de Chile; Rafael A. Burgos, DVM, MSc, Study Director — Universidad Austral de Chile; Juan C. Bertoglio, MD, Principal Investigator — Universidad Austral de Chile
Locations (2):
- Chile (2):
  - HOSPITAL REGIONAL de OSORNO, Osorno, Los Lagos Region
  - Hospital Clínico Regional, Valdivia, Los Ríos Region

IPD SHARING:
Plan to Share IPD: Yes
All these data has been accepted for publication in Clinical Rheumatology

REFERENCES:
- [Background] Agrawal S, Kandimalla ER. Antisense and/or immunostimulatory oligonucleotide therapeutics. Curr Cancer Drug Targets. 2001 Nov;1(3):197-209. doi: 10.2174/1568009013334160. PMID 12188879
- [Background] Clark W, Jobanputra P, Barton P, Burls A. The clinical and cost-effectiveness of anakinra for the treatment of rheumatoid arthritis in adults: a systematic review and economic analysis. Health Technol Assess. 2004 May;8(18):iii-iv, ix-x, 1-105. doi: 10.3310/hta8180. PMID 15130461
- [Background] FitzGerald GA, Patrono C. The coxibs, selective inhibitors of cyclooxygenase-2. N Engl J Med. 2001 Aug 9;345(6):433-42. doi: 10.1056/NEJM200108093450607. No abstract available. PMID 11496855
- [Background] Hidalgo MA, Romero A, Figueroa J, Cortes P, Concha II, Hancke JL, Burgos RA. Andrographolide interferes with binding of nuclear factor-kappaB to DNA in HL-60-derived neutrophilic cells. Br J Pharmacol. 2005 Mar;144(5):680-6. doi: 10.1038/sj.bjp.0706105. PMID 15678086
- [Background] Hengge UR, Brockmeyer NH, Goos M. Granulocyte colony-stimulating factor treatment in AIDS patients. Clin Investig. 1992 Oct;70(10):922-6. doi: 10.1007/BF00180439. PMID 1280496
- [Background] Iruretagoyena MI, Tobar JA, Gonzalez PA, Sepulveda SE, Figueroa CA, Burgos RA, Hancke JL, Kalergis AM. Andrographolide interferes with T cell activation and reduces experimental autoimmune encephalomyelitis in the mouse. J Pharmacol Exp Ther. 2005 Jan;312(1):366-72. doi: 10.1124/jpet.104.072512. Epub 2004 Aug 26. PMID 15331658
- [Background] Olsen NJ, Stein CM. New drugs for rheumatoid arthritis. N Engl J Med. 2004 May 20;350(21):2167-79. doi: 10.1056/NEJMra032906. No abstract available. PMID 15152062
- [Background] Setoguchi K, Misaki Y, Terauchi Y, Yamauchi T, Kawahata K, Kadowaki T, Yamamoto K. Peroxisome proliferator-activated receptor-gamma haploinsufficiency enhances B cell proliferative responses and exacerbates experimentally induced arthritis. J Clin Invest. 2001 Dec;108(11):1667-75. doi: 10.1172/JCI13202. PMID 11733562
- [Background] Smolen JS, Steiner G. Therapeutic strategies for rheumatoid arthritis. Nat Rev Drug Discov. 2003 Jun;2(6):473-88. doi: 10.1038/nrd1109. PMID 12776222
- [Background] Topol EJ. Failing the public health--rofecoxib, Merck, and the FDA. N Engl J Med. 2004 Oct 21;351(17):1707-9. doi: 10.1056/NEJMp048286. Epub 2004 Oct 6. No abstract available. PMID 15470193
- [Background] Yamamoto Y, Gaynor RB. Therapeutic potential of inhibition of the NF-kappaB pathway in the treatment of inflammation and cancer. J Clin Invest. 2001 Jan;107(2):135-42. doi: 10.1172/JCI11914. No abstract available. PMID 11160126
- [Background] Yazici Y, Erkan D, Paget SA. Monitoring by rheumatologists for methotrexate-, etanercept-, infliximab-, and anakinra-associated adverse events. Arthritis Rheum. 2003 Oct;48(10):2769-72. doi: 10.1002/art.11277. PMID 14558081
- [Background] Yazici Y, Erkan D, Paget SA. Monitoring methotrexate hepatic toxicity in rheumatoid arthritis: is it time to update the guidelines? J Rheumatol. 2002 Aug;29(8):1586-9. No abstract available. PMID 12180713
- [Result] Burgos RA, Hancke JL, Bertoglio JC, Aguirre V, Arriagada S, Calvo M, Caceres DD. Efficacy of an Andrographis paniculata composition for the relief of rheumatoid arthritis symptoms: a prospective randomized placebo-controlled trial. Clin Rheumatol. 2009 Aug;28(8):931-46. doi: 10.1007/s10067-009-1180-5. Epub 2009 Apr 29. PMID 19408036
- See also: Government of Chile - Science and Technology Development Fund (Study main sponsor) — http://www.fondef.cl